CLINICAL TRIAL: NCT06574282
Title: The COHIR Multi-center Study - a Non-interventional, Prospective, Multi-center Investigation With Exploratory Data Analysis to Assess the Proportion of Patients With Hypophosphatasia Presenting at the Department of Rheumatology and Establishment of an Algorithm to HPP Diagnosis.
Brief Title: Characteristics of Hypophosphatasia in Adult Patients in Rheumatology and Their Value in Developing an Algorithm to HPP-diagnosis - the COHIR Multi-center Study
Acronym: COHIRnational
Status: Recruiting | Type: Observational
Sponsor: University of Bonn (Other)
Responsible Party: Principal Investigator, Valentin Schäfer, Univ.-Prof. Dr. med. MuDr., University of Bonn
Other Study IDs: MED2-202002
Record Dates: First submitted 2024-08-25; First posted 2024-08-27 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Hypophosphatasia
Keywords: Hypophosphatasia; Hypophosphatasemia; Musculoskeletal complaints; Genetic disorder; Rare disease; Alkaline phosphatase gene; ALP; ALPL gene; Rheumatology; COHIR study; COHIR multi-center study; COHIRnational study; Prevalence; Diagnostic Algorithm; Metabolic bone diseases
MeSH Terms: conditions — Hypophosphatasia; Genetic Diseases, Inborn; Rare Diseases; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Persistant hypophosphatasemia
  Interventions: Diagnostic Test: Second alkaline phosphatase measurement
- Transient hypophosphatasemia (Control group without hypophosphatasia)
  Interventions: Diagnostic Test: Second alkaline phosphatase measurement

INTERVENTIONS:
Diagnostic Test: Second alkaline phosphatase measurement — (1-4 weeks after the 1st measurement)

SUMMARY:
Non-interventional, prospective, multi-center investigation with exploratory data analysis to assess the proportion of patients with hypophosphatasia presenting at departments of rheumatology and to establish an algorithm to HPP diagnosis

DETAILED DESCRIPTION:
Acronym: Expansion:

HPP =Hypophosphatasia COHIR ="Characteristics of Hypophosphatasia in Adult Patients in Rheumatology" ALPL =Alkaline Phosphatase

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age > 18 years
* Clinical suspicion of hypophosphatasia
* Evidence of an abnormal ALP (ALP below LLN) within the clinical routine screening

Exclusion Criteria:

* Failure to meet the inclusion criteria listed above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult patient presenting at the participating study site's rheumatology department with musculoskeletal complaints within the timeframe of the study conduct.
Sampling Method: Probability Sample
Enrollment: 720 (Estimated)
Dates: Start 2024-08-25 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of hypophosphatasia in adult patients in rheumatology | 36 months
  The primary aim of this prospective observational study is to determine the prevalence of hypophosphatasia in adult patients presenting with musculoskeletal symptoms in rheumatology.

CONTACTS AND LOCATIONS:
Overall Officials: Valentin S. Schäfer, Univ.-Prof. Dr. med. MUDr., Principal Investigator — University Hospital of Bonn
Locations (1):
- Clinic of Internal Medicine III, Department of Oncology, Haematology, Rheumatology and Clinical Immunology, University Hospital Bonn, Bonn, North Rhine-Westphali, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable request